CLINICAL TRIAL: NCT04640259
Title: This is a 100% Virtual (Remote) Study (Survey, and Voluntary Blood Donation) to Explore Potential Environmental, Lifestyle and Genetic Factors That May be Associated With Driver Mutations of Young Lung Cancer in the USA.
Brief Title: Epidemiology of Young Lung Cancer - Survey
Acronym: EoYLC
Status: Active, not recruiting | Type: Observational
Sponsor: Addario Lung Cancer Medical Institute (Other)
Collaborators: University of Southern California (Other); Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ALCMI-004
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- EGFR
  Interventions: Other: Online Survey
- ROS1
  Interventions: Other: Online Survey
- ALK
  Interventions: Other: Online Survey
- KRAS
  Interventions: Other: Online Survey
- NSCLC Other
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — Epidemiological Survey (approx 200 questions)

SUMMARY:
This is a 100% virtual (remote), case-case study to explore potential environmental, lifestyle and genetic factors that may be associated with driver mutations of young lung cancer in the U.S.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years and over; or the age of majority for their residential state at the time of enrollment
2. Documentation of primary NSCLC, any stage
3. Less than 50 years of age at the time of NSCLC diagnosis
4. Documentation of testing by a CLIA certified lab for genomic drivers of lung cancer
5. Willingness to undergo all study procedure
6. Provision of written informed consent

Exclusion Criteria:

1. Male or female aged less than 18 years; or less than the age of majority for their residential state
2. Greater than or equal to 50 years of age at the time of NSCLC diagnosis
3. No documentation of mutation testing
4. Unwilling to undergo all study procedures
5. Unable or unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 250 subjects distributed with at least 50 subjects among the most common driver mutation groups will be enrolled into the study:
  1. EGFR (del19 and L858R) - 50 subjects
  2. ROS1 - 50 subjects
  3. ALK - 50 subjects
  4. KRAS - 50 subjects
  5. Other Groups:
     1. Uncommon activating mutation for which specific targeted therapy exists (RET fusion, NTRK fusion, BRAF V600E, MET Exon14 skipping mutations, other activating EGFR mutations) - 25 subjects
     2. Non-targetable other mutations (p53, NF1, ATM, PIK3CA, RB, non-V600E BRAF, NTRK mutation) or no identified mutation. - 25 subjects Subjects with more than one mutation will be included.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Exploratory epidemiology correlates | 1 month
  Exploratory correlations between all questionnaire variables (demographic factors, medical history, smoking history, early life exposures (child and mother), residential history, occupational history, menstrual and reproductive history, diet, and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Nieva, MD, Principal Investigator — University of Southern California; Barbara Gitlitz, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - USC Keck School of Medicine, Los Angeles, California
  - Addario Lung Cancer Medical Institute, San Carlos, California

IPD SHARING:
Plan to Share IPD: No